CLINICAL TRIAL: NCT06372444
Title: Mechanisms of Acute Kidney Injury in Severe Infections
Acronym: PET-AKI
Status: Recruiting | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Miklos Lipcsey, Professor, Uppsala University Hospital
Other Study IDs: 995725
Record Dates: First submitted 2024-03-25; First posted 2024-04-18 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Sepsis; AKI - Acute Kidney Injury; Positron Emission Tomography (PET)
MeSH Terms: conditions — Sepsis; Acute Kidney Injury | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with sepsis and AKI
  Interventions: Radiation: Positron emission tomography (PET)
- Healthy controls
  Interventions: Radiation: Positron emission tomography (PET)

INTERVENTIONS:
Radiation: Positron emission tomography (PET) — Assessment of blood flow with marked water and assessment of neutrophil presence with neutrophil elastase tracer + CT

SUMMARY:
Renal perfusion and neutrophil-mediated inflammation will be assessed in the kidney in sepsis patients with acute kidney injury using positron emission tomography. For marked water will be used for renal perfusion and a newly developed PET tracer molecule (11C-GW457427) with specific binding to neutrophil elastase which provides a measure of the amount of infiltrating neutrophils in the renal parenchyma for inflammation. The study is performed in a PET-CT camera where anatomical imaging takes place at the same time as the PET examinations.

DETAILED DESCRIPTION:
To study renal perfusion and neutrophil-mediated inflammation 10 critically ill patients with sepsis and acute kidney injury (AKI) and 5 healthy volunteers as controls will be recruited and examined at one time with marked water followed by neutrophil elastase tracer. At the same time, a CT scan is performed for anatomy. Plasma levels of inflammatory mediators will be measured. Clinical data will be collected. The endpoints are changes in renal perfusion and increased presence of neutrophil elastase in the renal parenchyma.

ELIGIBILITY:
Inclusion Criteria:

Patients with sepsis and AKI

* > 30 years
* At least AKI stage 1 according to KDIGO where the last plasma creatinine is measured within 24 hours of the examination

Healthy volunteers

* > 30 years
* No previously known kidney disease
* Normal plasma creatinine value

Exclusion Criteria:

* Chronic renal failure (CKD stage >3a) or dialysis
* Instability in vital functions that makes PET-CT examination unsuitable
* Claustrophobia or other reasons that make the patient unable to lie still during the examination.
* Pregnancy and breastfeeding

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with sepsis and AKI and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-03 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Renal perfusion in patients with sepsis and acute kidney injury (AKI) measured by 15O-labeled water in dynamic positron emission tomography (PET) | PET performed within 10 days of AKI
  vs controls
Presence of neutrophil elastase in the kidneys in patients with sepsis and acute kidney injury (AKI) by 11C-GW457427 measured with dynamic positron emission tomography (PET) | PET performed within days of AKI
  vs controls

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala university hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
The underlying data for this study will not be made publicly available. However, the data may be acquired from the authors upon reasonable request after permission from the Swedish ethical review authority and under the limitations of the general data protection act of the European Union.